CLINICAL TRIAL: NCT04390906
Title: A Prospective Pilot Study of Cognitive Changes in Patients Receiving Partial Brain Radiation: Development of a Radiation Dose-toxicity Model for Neuroanatomic Targets
Brief Title: A Study of Cognitive Changes in Patients Receiving Brain Radiation
Status: Active, not recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Schmitt Program on Integrative Neuroscience (Unknown)
Responsible Party: Principal Investigator, Sara J Hardy, Resident, University of Rochester
Other Study IDs: RSRB00070001
Record Dates: First submitted 2020-04-10; First posted 2020-05-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Brain Tumor Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All participants: Participants will receive standard of care partial brain radiation therapy at discretion of their radiation oncologist

SUMMARY:
Cranial radiation therapy (RT), commonly used to treat benign and malignant brain tumors, can lead to cognitive impairments in domains not related to neuroanatomic structures directly impacted by the tumor. The study will prospectively enroll 75 patients with benign and low-grade brain tumors who will undergo partial brain RT, with either conventionally fractionated or hypofractionated schedules. Subjects will receive MRI scans at baseline, 6 months, and 12 months. Given the role of the limbic system in key cognitive functions affected by RT, researchers have a particular interest in characterizing MRI changes in the limbic system and thalamus in relation to memory and related processes.

Specific Aims:

1. To examine objective neurocognitive changes over time. The investigators hypothesize that they will see RT-induced neurocognitive impairment in up to 50% of patients after cranial RT.
2. To examine changes in brain tissue (via MRI) induced by off-target RT in patients with benign and low-grade brain tumors. The investigators specifically hypothesize that comapping of RT dose and MRI changes in the thalamus and limbic system (i.e., thalamic nuclei, hippocampus, fornix, hypothalamus/mammillary bodies, limbic lobe, cingulum) will be most distorted by off-target RT.
3. To examine the relationship between MRI changes for key neuroanatomic structures identified in Aim 1 with objective neurocognitive testing. The investigators hypothesize that cognitive decline will be correlated with damage revealed by MRI to limbic and thalamic structures.

This research will help to define which neuroanatomic structures are most at risk from RT-induced damage and will help ultimately establish new dose constraint guidelines for important structures to improve cognitive outcomes.

DETAILED DESCRIPTION:
Cranial radiation therapy (RT), commonly used to treat benign and malignant brain tumors, can lead to cognitive impairments in domains not related to neuroanatomic structures directly impacted by the tumor. This suggests that off-target RT, even at low doses, may have a negative cognitive impact by affecting neuroanatomic targets proximal or distal to the tumor. While constraints to minimize brain necrosis, ototoxicity, and optic neuropathy are well-established, RT dose tolerances for cognitive changes in key domains (memory, attention, executive function, and processing speed) that occur in RT-treated patients are poorly characterized. There is accumulating evidence that consideration of neuroanatomic targets could better explain cranial RT-mediated cognitive change. Additionally, a recent cooperative group phase III trial has shown that conformal avoidance of the hippocampus with whole brain RT can reduce cognitive impairment. Unfortunately, 60% of patients still had cognitive impairment at 6 months even with hippocampal avoidance, implying that other structures and networks are involved in cognitive deficits from RT and efforts to identify those structures are warranted. A major obstacle in the field has been difficulty identifying sites of off-target tissue damage that could impact cognition after RT. Given the role of the limbic system in key cognitive functions affected by RT, the investigators have a particular interest in characterizing changes in limbic system and thalamus in relation to memory and related processes.

The investigators plan to examine RT effects on neuroanatomic structures in the limbic system and thalamus as well as candidate structures identified systematically using magnetic resonance imaging (MRI). The investigators propose to prospectively enroll 75 patients with benign and low-grade brain tumors who will undergo partial brain RT, either conventionally fractionated or hypofractionated.

Neurocognitive testing will be obtained at baseline, 3, 6, and 12 months after RT using a battery of tests to assess visual and verbal memory, attention, executive function, and processing speed. Brain MRI, including high resolution T1 images, diffusion tensor imaging (DTI), and resting functional MRI (fMRI) sequences, will be evaluated at baseline, 6, and 12 months after RT.

This pilot study will provide preliminary data to identify key areas impacted by RT that can be followed up in future research.

Aim 1: To examine objective neurocognitive changes over time. Based on prior data, the investigators hypothesize that they will see RT-induced neurocognitive impairment in up to 50% of patients after cranial RT. The investigators will evaluate neurocognitive testing changes in the HVLT-R delayed recall (verbal memory) as their primary endpoint. As a secondary endpoint, they will evaluate a composite global deficit z-score as well as changes in cognitive domains of visual memory, attention, executive function and processing speed.

Aim 2: To examine changes in brain tissue (via MRI) induced by off-target RT in patients with benign and low-grade brain tumors. The investigators hypothesize that a detailed brain tissue injury mapping of off-target RT doses from pre to post-RT and reconstructed structural and functional connectivity (DTI and fMRI) will provide data on the relationship between RT dose and MRI changes in specific structures. The investigators specifically hypothesize that co-mapping of RT dose and MRI changes in the thalamus and limbic system (i.e., thalamic nuclei, hippocampus, fornix, hypothalamus/mammillary bodies, limbic lobe, cingulum) will be most distorted by off-target RT.

Aim 3: To examine the relationship between MRI changes for key neuroanatomic structures with neurocognitive testing. The investigators hypothesize that RT will impact several neuronal networks sub-serving multiple cognitive domains and cognitive decline (Aim 2) will be correlated with damage revealed by MRI to limbic and thalamic structures (Aim 1). This approach will allow identification of brain structures most associated with domain-specific cognitive impairment.

There is critical need for well-designed longitudinal studies that examine the impact of RT on neuroanatomic structures. Many of the studies that evaluate cognition with RT do not take into account neuroanatomic dose distributions. Even within the literature that evaluates neuroanatomic targets, there has not been a systematic approach to evaluation of neuroanatomic targets by RT. This research will help to define which neuroanatomic structures are most at risk from RT-induced damage and will help ultimately establish new dose constraint guidelines for important structures to improve cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old patients with brain tumors including low grade gliomas, meningiomas, acoustic neuromas, pituitary adenomas, craniopharyngiomas, hemangiopericytomas, pineal tumors, and other benign or slow-growing brain tumors
* Pathologic diagnosis will be required for gliomas, but not for other tumor types (though it will be recorded if available)
* Within 3 months prior to registration, patients must have a post gadolinium contrast-enhanced three dimensional spoiled gradient (SPGR), magnetization-prepared rapid gradient echo (MP-RAGE), or turbo field echo (TFE) MRI scan and an axial T2/FLAIR sequence. To yield acceptable image quality with the smallest possible axial slice thickness, , the imaging protocol should include the standard brain tumor protocol sequences: long DTI, sagittal SPGR, and brainlab sequences, resting functional MRI or their equivalent.
* Patients will need to be planned to receive fractionated radiation therapy or stereotactic radiation therapy, either fractionated or single fraction (enrollment must occur prior to radiation therapy so that baseline neurocognitive evaluation can be done)
* Surgical excision and/or chemotherapy treatment prior to enrollment is allowed
* Concurrent chemotherapy with radiation is allowed
* Antiepileptic drugs use, seizures, steroids, anticholinergic medications will be recorded but patients will not be excluded
* Hydrocephalus will be recorded, but patients will not be excluded

Exclusion Criteria:

* Prior cranial radiation therapy
* Other active malignancy
* Contraindication to MRI imaging such as implanted metal devices or foreign bodies
* Contraindication to gadolinium contrast administration during MR imaging such as allergy or insufficient renal function
* Intractable seizures while on adequate anticonvulsant therapy-more than 1 seizure per month for the past 2 months
* Life expectancy <6 months due to other severe comorbidity
* Due to limitations in our ability to test patients in languages other than English, patients will have to be English-speaking
* Diagnosis of pre-existing dementia (clinically significant as defined by a neurologist or other provider), neurodegenerative, or neuro-inflammatory conditions as made by an appropriate health care professional such as a neurologist
* Inability to participate in neuro-cognitive testing
* Significant aphasia leading to difficulty participating in neuro-cognitive testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low grade or benign brain tumors planned to receive partial brain radiation.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change on HVLT-R delayed recall | baseline to 6 months
  Serial neurocognitive testing using raw scores from the HVLT-R delayed recall

SECONDARY OUTCOMES:
Correlation of change in fractional anisotropy (FA) on diffusion tensor imaging (DTI) in the thalamus and limbic system with RT dose | baseline to 6 months
  Correlation of longitudinal change in FA for limbic system white matter regions of interest and RT dose
Correlation of change in mean diffusivity (MD) on diffusion tensor imaging (DTI) in the thalamus and limbic system with RT dose | baseline to 6 months
  Correlation of longitudinal change in MD for limbic system white matter regions of interest and RT dose
Correlation of change on resting state functional MRI (rs-fMRI) and RT dose | baseline to 6 months
  Correlation of longitudinal change in connectivity measures for limbic system/thalamus regions of interest on rs-fMRI and RT dose
Correlation of change in region of interest volumes and RT Dose | baseline to 6 months
  Correlation of longitudinal change in volume for gray matter limbic system structures/thalamus on T1 MRI and RT dose
Change in global cognitive function | baseline to 6 months
  Serial neurocognitive testing using scores from the HVLT-R, BVMT-R, CTMT, COWA, DMS, PAL, ERT, SWM. Results from these tests will be combined into a composite global cognition z-score [-3 to +3]

CONTACTS AND LOCATIONS:
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hardy SJ, Finkelstein AJ, Tivarus M, Culakova E, Mohile N, Weber M, Lin E, Zhong J, Usuki K, Schifitto G, Milano M, Janelsins-Benton MC. Cognitive and neuroimaging outcomes in individuals with benign and low-grade brain tumours receiving radiotherapy: a protocol for a prospective cohort study. BMJ Open. 2023 Feb 15;13(2):e066458. doi: 10.1136/bmjopen-2022-066458. PMID 36792323